CLINICAL TRIAL: NCT05794763
Title: The Body Project: Comparing the Effectiveness of an In-person and Virtually Delivered Intervention.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Eric Stice, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 64138
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Eating Disorders
Keywords: Prevention; Peer Leader; Feeding and Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor at the 3-month follow-up is blind to participant randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Project: In Person Delivery (Experimental): In the in-person peer-led group intervention, participants voluntarily engage in verbal, written, and behavioral exercises in which they critique and discuss the costs of pursuing the thin-ideal ideal. The intervention is 4 sessions long (1-hr each) and is administered by trained peer facilitators who use an intervention script. Participants will be asked to complete weekly home exercises throughout the course of the intervention.
  Interventions: Behavioral: Peer Led Group Intervention
- Body Project: Virtual Delivery (Experimental): In the virtual peer-led group intervention held over Zoom, participants voluntarily engage in verbal, written, and behavioral exercises in which they critique and discuss the costs of pursuing the thin-ideal ideal. The intervention is 4 sessions long (1-hr each) and is administered by trained peer facilitators who use an intervention script. Participants will be asked to complete weekly home exercises throughout the course of the intervention.
  Interventions: Behavioral: Peer Led Group Intervention

INTERVENTIONS:
Behavioral: Peer Led Group Intervention — A four-week dissonance-based program where individuals with body image concerns complete verbal, written, and behavioral activities. The program consists of four 60-minute sessions
  Other Names: Body Project

SUMMARY:
This present study will compare the efficacy of in-person versus virtually-delivered Body Project groups. It will also evaluate whether this body acceptance class produces greater reductions in eating disorder risk factor symptoms (pursuit of the thin ideal, body dissatisfaction, dieting, dietary restraint, negative affect, eating disorder symptoms, and the future onset of eating disorders over a 3-month follow-up in this population. It will also evaluate the effectiveness of this body acceptance class's ability to impact social appearance anxiety, body compassion, and self-stigma surrounding attaining help.

DETAILED DESCRIPTION:
Dozens of eating disorder prevention programs have been evaluated, but only the 4-hr Body Project has reduced eating disorder symptoms and future eating disorder onset over 3-4 year follow-up, produced larger reductions in outcomes than credible alternative interventions, been shown to engage the intervention target (valuation of the thin beauty ideal), and produced effects in trials from several independent teams. The proposed study will evaluate the effectiveness of a peer-implemented, virtually delivered, body acceptance class compared to a peer-implemented, in-person delivery of the same class. Participation in the intervention will last four weeks. Participants will be randomly assigned to the in-person or virtual body acceptance class. Assessments will take place at pre-intervention, post-intervention, and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria: Participants had to express body image concerns and all gender identities besides cisgender and transgender men were eligible.

Exclusion Criteria:

* Cisgender and transgender men were excluded due to the fact that The Body Project is typically administered with groups of all cisgender women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All gender identities besides cisgender and transgender men were eligible.
Enrollment: 69 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - St. Mary's College of Maryland, Saint Marys City, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Body Project: In Person Delivery | Body Project: Virtual Delivery
Started | 33 | 36
Completed | 33 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Body Project: In Person Delivery | Body Project: Virtual Delivery | Total
Number analyzed (Participants) | 33 | 36 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 6 | 13
  Between 18 and 65 years | 26 | 30 | 56
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 22 | 22 | 44
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 33 | 36 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change Over Time in Body Dissatisfaction
Description: Ten items from the Satisfaction and Dissatisfaction with Body Parts Scale assessed satisfaction with body parts with a response scale ranging from 1 = extremely dissatisfied to 6 = extremely satisfied. The mean score across the items is reported. Overall scores can range from 1 to 6 and a higher score indicate a greater level of body satisfaction.
Time Frame: Pre intervention obtained on intake, and immediately post intervention (after completion of 4 weeks of group session once a week)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Body Project: In Person Delivery | Body Project: Virtual Delivery
Number analyzed (Participants) | 33 | 36
score on a scale | .42 [0.1359 to 0.7241] | 0.51 [0.3329 to 0.6871]

2. Primary Outcome: Change Over Time in Thin Ideal Internalization
Description: The eight-item Ideal-Body Stereotype Scale-Revised will assess endorsement of the thin beauty ideal using a response scale ranging from 1 = strongly disagree to 5 = strongly agree. The mean score across the items is reported. Overall scores can range from 1 to 5 and a higher score indicates a greater level of thin ideal internalization.
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: scale
Arm/Group | Body Project: In Person Delivery | Body Project: Virtual Delivery
Number analyzed (Participants) | 33 | 36
scale | -0.64 [-1.0115 to -0.2685] | -0.59 [-0.9544 to -0.2256]

3. Secondary Outcome: Change Over Time in Negative Affect
Description: Twenty items from the sadness, guilt, and fear/anxiety subscales from the Positive Affect and Negative Affect Scale-Revised will assess negative affect. Participants reported the extent to which they had felt negative emotions on scales ranging from 1 = very slightly or not at all to 5 = extremely. The mean score across the items is reported. Overall scores can range from 1 to 5 and a higher score indicates a greater level of negative affect.
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: scale score
Arm/Group | Body Project: In Person Delivery | Body Project: Virtual Delivery
Number analyzed (Participants) | 33 | 36
scale score | -0.17 [-0.64 to 0.30] | -0.41 [-0.8023 to -0.0177]

4. Secondary Outcome: Change Over Time in Dieting
Description: The 10-item Dutch Restrained Eating Scale will assess the frequency of dieting behaviors using a response scale ranging from 1 = never to 5 = always. The mean score across the items is reported. Overall scores can range from 1 to 5 and a higher score indicates greater frequency of dieting behaviors.
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: scale score
Arm/Group | Body Project: In Person Delivery | Body Project: Virtual Delivery
Number analyzed (Participants) | 33 | 36
scale score | -0.48 [-0.9445 to -0.0155] | -0.77 [-1.137 to -0.403]

5. Secondary Outcome: Body Comparison Orientation
Description: The six selected items from the Body, Eating, and Exercise Comparison Orientation Scale will assess the frequency of body comparisons using a response scale ranging from 1 = strongly disagree to 5 = strongly agree. The mean score across the items is reported. Overall scores can range from 1 to 5 and a higher score indicates greater frequency of body comparison.
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: scale score
Arm/Group | Body Project: In Person Delivery | Body Project: Virtual Delivery
Number analyzed (Participants) | 33 | 36
scale score | -0.38 [-0.8272 to 0.0672] | -0.60 [-1.0454 to -0.1546]

6. Secondary Outcome: Change Over Time in Social Appearance Anxiety
Description: The 16-item Social Appearance Anxiety Scale will assess levels of social appearance anxiety using a response scale ranging from 1 = not at all to 5 = extremely.
Time Frame: Pre intervention obtained on intake, and immediately post intervention.
Reporting Status: Not Posted

7. Secondary Outcome: Change Over Time in Body Compassion
Description: The 10-item Body Appreciation Scale-2 will assess levels of body compassion using a response scale ranging from 1 = never to 5 = always.
Time Frame: Pre intervention obtained on intake, and immediately post intervention.
Reporting Status: Not Posted

8. Secondary Outcome: Change Over Time in Self-Stigma of Seeking Help Scale
Description: The 10-item Self-Stigma of Seeking Help Scale will assess participants' views towards seeking help using a scale ranging from 1 = strongly disagree to 5 = strongly agree.
Time Frame: Pre intervention obtained on intake, and immediately post intervention.
Reporting Status: Not Posted

9. Secondary Outcome: Number of Eating Disorder Behaviors (Events) as a Measure of Change Over Time in Eating Disorder Symptoms
Description: Interviewer assesses frequency of eating disorder behaviors using Eating Disorder Diagnostic Interview.
Time Frame: Pre intervention and 3 months after the end of the intervention.
Measure: Mean (95% Confidence Interval); unit: events
Arm/Group | Body Project: In Person Delivery | Body Project: Virtual Delivery
Number analyzed (Participants) | 33 | 36
events | -5.22 [-11.225 to 0.7852] | -3.68 [-9.0126 to 1.6526]

10. Secondary Outcome: Body Project Specific Attitude Measures
Description: 7 items assessing attitudes that are targeted as part of The Body Project training using a response scale ranging from 1 = strongly disagree to 5 = strongly agree.
Time Frame: Pre intervention obtained on intake, and immediately post intervention.
Reporting Status: Not Posted

11. Secondary Outcome: Body Project Specific Outcome Measures
Description: as for outcome 10
Time Frame: Pre intervention obtained on intake, and immediately post intervention.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4-week intervention period plus 3-month follow-up
Arm/Group | Body Project: In Person Delivery | Body Project: Virtual Delivery
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/36
Other Adverse Events (participants affected / at risk) | 0/33 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT05794763/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT05794763/SAP_001.pdf
  • Informed Consent Form (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT05794763/ICF_002.pdf